CLINICAL TRIAL: NCT03724890
Title: A Multicenter, Open-Label, Dose Escalation Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of the DNA-PK Inhibitor M3814 in Combination With Avelumab With and Without Palliative Radiotherapy in Participants With Selected Advanced Solid Tumors
Brief Title: Study of Avelumab-M3814 Combinations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS201964_0001
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Oncology; Solid Tumors
Keywords: Palliative Radiotherapy; Advanced solid tumors; M3814; Avelumab
MeSH Terms: conditions — Neoplasms | interventions — peposertib; avelumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: M3814 + Avelumab (Experimental)
  Interventions: Drug: M3814; Drug: Avelumab
- Part B: M3814 + Avelumab + Radiotherapy (RT) (Experimental)
  Interventions: Drug: M3814; Drug: Avelumab; Radiation: Radiotherapy
- Part FE: M3814 + Avelumab (fasted/fed state) (Experimental)
  Interventions: Drug: M3814; Drug: Avelumab

INTERVENTIONS:
Drug: M3814 — Participants received M3814 twice daily (BID) continuously starting from Day 1 until progressive disease (PD) or unacceptable toxicity.
  Other Names: Peposertib; MSC2490484A
  Arms: Part A: M3814 + Avelumab; Part FE: M3814 + Avelumab (fasted/fed state)
Drug: M3814 — Participants received M3814 concomitantly with RT once (QD) daily starting Day 1 for 5 days per week for 2 weeks in total.
  Other Names: Peposertib; MSC2490484A
  Arms: Part B: M3814 + Avelumab + Radiotherapy (RT)
Drug: Avelumab — Participants received avelumab once every 2 weeks (Q2W) starting from Day 1 until PD or unacceptable toxicity.
Radiation: Radiotherapy — Participants received radiotherapy at the dose of 3 grays (Gy) per day starting Day 1 for 5 days per week for 2 weeks.
  Arms: Part B: M3814 + Avelumab + Radiotherapy (RT)

SUMMARY:
The main purpose of the study was to evaluate a safe, tolerable recommended Phase II dose (RP2D) and/or the maximum tolerated dose (MTD) of M3814 when given in combination with avelumab with and without radiotherapy in participants with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Part A and Part FE (M3814 + avelumab): Participants had histologically or cytologically proven advanced or metastatic solid tumors for which no standard therapy exists, standard therapy has failed, or participants are intolerant to or have rejected established therapy known to provide clinical benefit for their condition
* Part B (M3814 + Radiotherapy [RT] + avelumab): histologically or cytologically proven advanced or metastatic solid tumors for which no standard therapy exists, standard therapy has failed, or participants are intolerant to or have rejected established therapy known to provide benefit for their condition and are amenable to receive RT
* Part A, B and FE: Measurable or evaluable disease according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v 1.1)
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 1 at study entry
* Part A, B and FE: Female participants of childbearing potential should be willing to use a highly effective contraceptive method
* Part A, B and FE: Male participants should agree to refrain from donating sperm plus, either: abstain from any activity that allows for exposure to ejaculate
* Use an adequate method of contraception starting with the first dose of study therapy through 90 days after the last dose of study therapy
* Part A, B and FE: Be willing to provide informed consent for the trial
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants who had received prior chemotherapy, hormonal anticancer therapy with the exception of luteinizing hormone-releasing hormone analogs, biologic therapy, or any other anticancer therapy within 28 days of the first dose of study treatments (6 weeks for nitrosoureas or mitomycin C)
* Participants who had undergone major surgery for any reason, except diagnostic biopsy, within 4 weeks of the study intervention and/or has not fully recovered from the surgery within 4 weeks of the study intervention
* Participants with evidence of active or history of autoimmune disease that might deteriorate when receiving an immune-stimulatory agent
* Participants with brain metastases, except those meeting the following criteria: a) brain metastases that have been treated locally and are clinically stable for greater than or equal to (>=) 4 weeks prior to randomization b) no ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable) c) participants must be either off steroids or on a stable or decreasing dose of less than (<) 10 milligrams (mg) daily prednisone (or equivalent)
* Participants with severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year), psychiatric or substance abuse disorders; or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study intervention administration or may interfere with the interpretation of study results
* Participants requiring systemic immunosuppressive agents (such as steroids) for any reason who cannot be tapered off these drugs before start of study intervention, with the following exceptions: a) participants with adrenal insufficiency, may continue corticosteroids at physiologic replacement dose, equivalent to less than or equal to (<=) 10 mg prednisone daily b) participants requiring steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intra-ocular, or inhalation) is permitted c) participants with previous or ongoing administration of systemic steroids for the management of an acute allergic phenomenon planned to be completed in 14 days, or that the dose after 14 days will be equivalent to <= 10 mg prednisone daily
* Participants with a history of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome, Hepatitis B virus or Hepatitis C and with history of infection must have a polymerase chain reaction (PCR) documentation that infection is cleared
* Participants who had received a live vaccine within 30 days prior to the first dose of trial treatment
* Participants with known prior severe hypersensitivity to any of the investigational products or any component in its formulations
* Participants with evidence of additional malignancy within the last 5 years unless a complete remission without further recurrence was achieved at least 2 years prior to study entry and participants were deemed to have been cured with no additional therapy required or anticipated to be required. Participants with treated nonmelanoma skin cancers, carcinoma in situ of skin, bladder, cervix, colon/rectum, breast, or prostate may participate
* Participants pretreated with immunotherapy who have, any history of dose limiting toxicities (DLTs) with prior immunotherapy agents, including Grade 3/4 immune-related adverse events (irAEs); irreversible irAEs; Grade greater than or equals to (>=) 3 irAEs that did not respond to steroid rescue; or neurologic irAE with significant clinical sequelae
* Participants with irAE requiring hormone replacement therapy (e.g., thyroxine, insulin, or physiologic dose of corticosteroid replacement therapy for adrenal or pituitary insufficiency) may participate as long as the endocrinopathy is well controlled and the participant is not otherwise symptomatic from hormone insufficiency
* Physiologic corticosteroid dose is defined as <= 10 mg daily of prednisone or equivalent
* for Part B only:
* Participants who had confirmed esophagitis and in whom radiation planning target volume will include any portion of the esophagus, the participant is not eligible unless an esophageal endoscopy rules out the presence of esophagitis
* Participants in whom more than 10 percent (%) of the total esophagus volume might receive more than 15 gray (Gy) (50% of the prescribed radiotherapy [RT] dose)
* Participants who have had previous radiotherapy to the same region as intended to be irradiated in this study within the past 12 months
* Participants who had had extensive previous radiotherapy on >= 30% of bone marrow reserve or prior bone marrow/stem cell transplantation within 5 years before study start
* If participant hepatic metastatic lesion is selected to be irradiated: - the non-tumor liver volume < 700 milli liters (mL); - Child-Pugh score >= 8
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (8):
- United States (8):
  - H. Lee Moffitt Cancer Center and Research Institute, Inc, Tampa, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - Mount Sinai - PRIME (10707), Lake Success, New York
  - UC Health Clinical Trials Office (10702), Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - Greenville Hospital System University Medical Center (ITOR), Greenville, South Carolina
  - Vanderbilt-Ingram Cancer Center (8867), Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- [Background] Perez B, Aljumaily R, Marron TU, Shafique MR, Burris H, Iams WT, Chmura SJ, Luke JJ, Edenfield W, Sohal D, Liao X, Boesler C, Machl A, Seebeck J, Becker A, Guenther B, Rodriguez-Gutierrez A, Antonia SJ. Phase I study of peposertib and avelumab with or without palliative radiotherapy in patients with advanced solid tumors. ESMO Open. 2024 Feb;9(2):102217. doi: 10.1016/j.esmoop.2023.102217. Epub 2024 Feb 5. PMID 38320431
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201964_0001
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant signed informed consent: 27-Nov-2018; Clinical data cutoff date: 05 Aug 2022
Pre-assignment Details: This study was conducted in 3 parts; Part A, Part B and Part Food Effect (FE). Participants who enrolled in Part A of study were not eligible to participate in Part B and Part FE.
Groups:
- Part A: M3814 100 mg BID + Avelumab 800 mg Q2W: Participants received 100 milligrams (mg) of M3814 orally twice daily (BID) along with 800 mg of Avelumab once every 2 weeks (Q2W) from Day 1 until progressive disease (PD) or unacceptable toxicity. M3814 will be administered without food.
- Part A: M3814 200 mg BID + Avelumab 800 mg Q2W: Participants received 200 mg of M3814 orally BID along with 800 mg of Avelumab Q2W from Day 1 until PD or unacceptable toxicity. M3814 will be administered without food.
- Part A: M3814 250 mg BID + Avelumab 800 mg Q2W: Participants received 250 mg of M3814 orally BID along with 800 mg of Avelumab Q2W from Day 1 until PD or unacceptable toxicity. M3814 will be administered without food.
- Part A: M3814 300 mg BID + Avelumab 800 mg Q2W: Participants received 300 mg of M3814 orally BID along with 800 mg of Avelumab Q2W from Day 1 until PD or unacceptable toxicity. M3814 will be administered without food.
- Part A: M3814 400 mg BID + Avelumab 800 mg Q2W: Participants received 400 mg of M3814 orally BID along with 800 mg of Avelumab Q2W from Day 1 until PD or unacceptable toxicity. M3814 will be administered without food.
- Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT: Participants received 100 mg of M3814 along with radiotherapy (RT) at 3 grays (Gy) once daily (QD) starting on Day 1 for 5 days per week for 2 weeks in combination with intravenous infusion of Avelumab at a dose of 800 mg Q2W starting from Day 1 until PD or unacceptable toxicity. M3814 will be administered without food.
- Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT: Participants received 150 mg of M3814 along with RT at 3 Gy QD starting on Day 1 for 5 days per week for 2 weeks in combination with intravenous infusion of Avelumab at a dose of 800 mg Q2W starting from Day 1 until PD or unacceptable toxicity. M3814 will be administered without food.
- Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT: Participants received 200 mg of M3814 along with RT at 3 Gy QD starting on Day 1 for 5 days per week for 2 weeks in combination with intravenous infusion of Avelumab at a dose of 800 mg Q2W starting from Day 1 until PD or unacceptable toxicity. M3814 will be administered without food.
- Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT: Participants received 250 mg of M3814 along with RT at 3 Gy QD starting on Day 1 for 5 days per week for 2 weeks in combination with intravenous infusion of Avelumab at a dose of 800 mg Q2W starting from Day 1 until PD or unacceptable toxicity. M3814 will be administered without food.
- Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W: Participants were administered 100 mg M3814 tablet orally BID in combination with i.v of avelumab at a dose of 800 mg Q2W throughout the whole study under fasted condition with the exception of fed condition on Day 1 and Day 22. The summary statistics for demographics, safety and efficacy is based on dose level but not fast/fed condition which is not fit for purpose.
- Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W: Participants were administered 200 mg M3814 tablet orally BID in combination with i.v of avelumab at a dose of 800 mg Q2W throughout the whole study under fasted condition with the exception of fed condition on Day 1 and Day 22. The summary statistics for demographics, safety and efficacy is based on dose level but not fast/fed condition which is not fit for purpose.
Period: Overall Study
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W
Started | 4 | 11 | 4 | 6 | 4 | 3 | 3 | 4 | 9 | 4 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 11 | 4 | 6 | 4 | 3 | 3 | 4 | 9 | 4 | 5
Not completed — Death | 2 | 6 | 3 | 5 | 2 | 0 | 2 | 3 | 4 | 2 | 2
Not completed — Lost to Follow-up | 0 | 3 | 0 | 1 | 2 | 2 | 1 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 1
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Full analysis set included all participants who receive at least one dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W | Total
Number analyzed (Participants) | 4 | 11 | 4 | 6 | 4 | 3 | 3 | 4 | 9 | 4 | 5 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59 (17.5) | 55 (19.6) | 53 (18.6) | 64 (4.1) | 53 (7.7) | 59 (17.3) | 69 (13.8) | 62 (7.2) | 61 (8.6) | 64 (9.3) | 68 (17.3) | 60 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 4 | 3 | 3 | 1 | 3 | 2 | 4 | 2 | 4 | 32
  Male | 4 | 5 | 0 | 3 | 1 | 2 | 0 | 2 | 5 | 2 | 1 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 4 | 10 | 4 | 6 | 4 | 2 | 3 | 4 | 8 | 4 | 5 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 5 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 11
  White | 3 | 6 | 3 | 6 | 2 | 2 | 3 | 3 | 8 | 4 | 4 | 44
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs) Assessed Using National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) Version 5.0
Description: A DLT was defined as any Grade more than or equal to >= 3 nonhematologic Adverse Event(AE) or any Grade>= 4 hematologic,, occurring during the DLT period that is related to any of the study interventions. In addition, a DLT is considered: Grade 3 thrombocytopenia with medically concerning bleeding, Any febrile neutropenia. A study intervention-related Treatment emergent Adverse Event(TEAE) is of potential clinical significance such that further dose escalation would expose participants to unacceptable risk. Any toxicity related to study intervention that causes the participant to receive less than 80% of M3814 during DLT period, evidence of study treatment-related hepatocellular injury for more than 3 days, such as> 5-fold elevations above the Upper Limits of Normal (ULN) of Alanine Aminotransferase (ALT) or Aspartate Aminotransferase(AST) with or without elevation of serum total bilirubin to > 2 × ULN. Number of Participants with DLT Grade >= 3 were reported.
Time Frame: Day 1 up to Day 21
Population: DLT analysis set included all participants who received at least 34 of 42 daily doses of M3814 and 2 administrations of avelumab during the DLT evaluation period and remained on study for the entirety of the DLT evaluation period, or participants who experienced a DLT during the DLT evaluation period and received any amount of any study intervention. The DLT evaluation period was defined as the first 21 days of the study, following the start of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 5 | 2 | 4 | 4
Participants | 0 | 0 | 1 | 1 | 3

2. Primary Outcome: Part B: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs) Assessed Using National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) Version 5.0
Description: as for outcome 1
Time Frame: Day 1 up to Day 28
Population: DLT analysis set included all participants who received 8 of 10 daily doses of peposertib, 8 fractions of radiotherapy, and 3 administrations of avelumab during the DLT evaluation period and remained on study for the entirety of the DLT evaluation period or participants who experienced a DLT during the DLT evaluation period and received any amount of any study intervention. The DLT evaluation period was defined as the first 28days of the study, following the start of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 3 | 3 | 3 | 4
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Part Food Effect (FE): Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero to 6 Hour (AUC0-6hour) of M3814
Description: Area under the plasma concentration versus time curve from time zero to 6 hours post dosing for M3814 was reported.
Time Frame: Pre-dose, 1, 2, 4 and 6 hours post-dose on Day 1; Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Day 15; Pre-dose, 2, 4 and 6 hours post-dose on Day 22
Population: The Pharmacokinetic (PK) Analysis Set included all subjects who received at least one administration of M3814 and avelumab and had at least one measurable post-dose PK sample. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 3 | 2
hour*nanogram per milliliter (h*ng/mL)
  Day 1: number analyzed (Participants) | 3 | 1
  Day 1 | 1520 (159.7) | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values
  Day 15 | 6250 (86.4) | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values
  Day 22: number analyzed (Participants) | 1 | 1
  Day 22 | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values

4. Primary Outcome: Part FE: Maximum Observed Plasma Concentration (Cmax) of M3814
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 3 | 5
nanogram per milliliter (ng/mL)
  Day 1 | 563 (100.5) | 950 (119.6)
  Day 15: number analyzed (Participants) | 3 | 2
  Day 15 | 1370 (63.2) | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values
  Day 22: number analyzed (Participants) | 3 | 1
  Day 22 | 1070 (99.4) | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values

5. Secondary Outcome: Part A: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-related TEAEs and Serious TEAEs According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Description: An Adverse Event(AE) is any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal relationship with this treatment. Therefore, an AE can be any unfavorable and unintended sign, symptom, or disease associated with the use of a medicinal product, regardless if it is considered related to the medicinal product. Serious AE: AE that resulted in death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE: AE with onset after start of treatment or with onset date before the treatment start date but worsening after treatment start date. TEAEs included both serious and non-serious TEAEs. Treatment-related TEAEs: reasonably related to study intervention. Number of participants with TEAEs, treatment related TEAEs and serious TEAEs were reported.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 516 days)
Population: Safety Analysis Set included all participants who received at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 11 | 4 | 6 | 4
Participants
  TEAEs | 3 | 11 | 4 | 6 | 4
  Related TEAE | 3 | 10 | 3 | 4 | 4
  Serious TEAE | 0 | 6 | 4 | 4 | 4

6. Secondary Outcome: Part B: Number of Participants With Treatment-Emergent Adverse Events, Treatment-related TEAEs and Serious TEAEs According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Description: as for outcome 5
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 513 Days)
Population: Safety Analysis Set included all participants who received at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 3 | 3 | 4 | 9
Participants
  TEAEs | 3 | 3 | 4 | 9
  Treatment-related TEAEs | 3 | 3 | 4 | 8
  Serious TEAEs | 2 | 1 | 1 | 6

7. Secondary Outcome: Part FE: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-related TEAEs and Serious TEAEs According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Description: as for outcome 5
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 404 Days)
Population: Safety Analysis Set included all participants who received at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 5
Participants
  TEAEs | 4 | 5
  Treatment-related TEAEs | 3 | 5
  Serious TEAEs | 2 | 3

8. Secondary Outcome: Part A: Number of Participants With Abnormalities Grade Greater Than or Equals to (>=) 3 in Laboratory Test Values
Description: The laboratory measurements included hematology and biochemistry values were graded with National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 toxicity grades (where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening and Grade 5 = death). Number of participants with abnormalities Grade >= 3 in laboratory test values were reported.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 516 days)
Population: Safety Analysis Set included all participants who received at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 11 | 4 | 6 | 4
Participants | 0 | 7 | 4 | 5 | 4

9. Secondary Outcome: Part B: Number of Participants With Abnormalities Grade Greater Than or Equals to (>=) 3 in Laboratory Test Values
Description: as for outcome 8
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 513 Days)
Population: Safety Analysis Set included all participants who received at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 3 | 3 | 4 | 9
Participants | 0 | 0 | 0 | 2

10. Secondary Outcome: Part FE: Number of Participants With Abnormalities Grade Greater Than or Equals to (>=) 3 in Laboratory Test Values
Description: as for outcome 8
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 404 Days)
Population: Safety Analysis Set included all participants who received at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

11. Secondary Outcome: Part A: Number of Participants With Clinically Meaningful Change From Baseline in Electrocardiogram (ECG)
Description: Number of participants with clinically meaningful change from baseline in ECG parameters were reported. Clinically Meaningful Change was decided by the investigator. The 12-lead ECGs were recorded after the participants have rested for at least 5 minutes in supine position. The parameters included heart rate (HR), Respiratory Rate, Pulse Rate, QRS, QT and QTcB calculated by the Bazett formula.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 516 days)
Population: Safety Analysis Set included all participants who received at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 11 | 4 | 6 | 4
Participants | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Part B: Number of Participants With Clinically Meaningful Change From Baseline in Electrocardiogram (ECG)
Description: as for outcome 11
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 513 Days)
Population: Safety Analysis Set included all participants who received at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 3 | 3 | 4 | 9
Participants | 0 | 0 | 0 | 0

13. Secondary Outcome: Part FE: Number of Participants With Clinically Meaningful Change From Baseline in Electrocardiogram (ECG)
Description: as for outcome 11
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 404 Days)
Population: Safety Analysis Set included all participants who received at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

14. Secondary Outcome: Part A: Number of Participants With Clinically Meaningful Change From Baseline in Vital Signs
Description: Number of participants with clinically meaningful change from baseline in vital signs. Clinically Meaningful Change was decided by the investigator. Vital signs included oral body temperature, systolic blood pressure, diastolic blood pressure, and pulse rate.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 516 days)
Population: Safety Analysis Set included all participants who received at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 11 | 4 | 6 | 4
Participants | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Part B: Number of Participants With Clinically Meaningful Change From Baseline in Vital Signs
Description: as for outcome 14
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 513 Days)
Population: Safety Analysis Set included all participants who received at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 3 | 3 | 4 | 9
Participants | 0 | 0 | 0 | 0

16. Secondary Outcome: Part FE: Number of Participants With Clinically Meaningful Change From Baseline in Vital Signs
Description: as for outcome 14
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 404 Days)
Population: Safety Analysis Set included all participants who received at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

17. Secondary Outcome: Part A: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance: Baseline Score Versus (Vs) Worst Post-baseline Score
Description: ECOG PS score is widely used by doctors and researchers to assess how a participants disease is progressing and is used to assess how the disease affects the daily living abilities of the participant and determine appropriate treatment and prognosis. The score ranges from Grade0 to Grade5, where Grade0=Fully active, able to carry on all pre-disease performance without restriction, Grade1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (like light house work, office work), Grade2 = Ambulatory and capable of all self-care but unable to carry out any work activities, Grade3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours and Grade4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair, Grade5=Death.ECOG performance status was reported in terms of number of participants with baseline value vs worst post-baseline value.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 516 days)
Population: Safety Analysis Set included all participants who receive at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 11 | 4 | 6 | 4
Participants
  Baseline score 0, worst post-baseline score 0 | 2 | 2 | 1 | 1 | 0
  Baseline score 0, worst post-baseline score 1 | 0 | 1 | 1 | 2 | 0
  Baseline score 0, worst post-baseline score 2 | 0 | 0 | 0 | 0 | 1
  Baseline score 0, worst post-baseline score 3 | 0 | 1 | 0 | 0 | 2
  Baseline score 0, worst post-baseline score 4 | 0 | 0 | 0 | 0 | 0
  Baseline score 0, worst post-baseline score 5 | 0 | 0 | 0 | 0 | 0
  Baseline score 0, worst post-baseline score Missing | 0 | 0 | 1 | 0 | 0
  Baseline score 1, worst post-baseline score 0 | 0 | 0 | 0 | 0 | 0
  Baseline score 1, worst post-baseline score 1 | 2 | 4 | 0 | 2 | 1
  Baseline score 1, worst post-baseline score 2 | 0 | 1 | 0 | 0 | 0
  Baseline score 1, worst post-baseline score 3 | 0 | 2 | 0 | 1 | 0
  Baseline score 1, worst post-baseline score 4 | 0 | 0 | 0 | 0 | 0
  Baseline score 1, worst post-baseline score 5 | 0 | 0 | 0 | 0 | 0
  Baseline score 1, worst post-baseline score Missing | 0 | 0 | 1 | 0 | 0

18. Secondary Outcome: Part B:Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance: Baseline Score Versus (Vs) Worst Post-baseline Score
Description: as for outcome 17
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 513 Days)
Population: Safety Analysis Set included all participants who received at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 3 | 3 | 4 | 9
Participants
  Baseline score 0, worst post-baseline score 0 | 1 | 0 | 0 | 2
  Baseline score 0, worst post-baseline score 1 | 1 | 2 | 3 | 1
  Baseline score 0, worst post-baseline score 2 | 0 | 0 | 0 | 1
  Baseline score 0, worst post-baseline score 3 | 0 | 0 | 0 | 0
  Baseline score 0, worst post-baseline score 4 | 0 | 0 | 0 | 0
  Baseline score 0, worst post-baseline score 5 | 0 | 0 | 0 | 0
  Baseline score 0, worst post-baseline score Missing | 0 | 0 | 0 | 0
  Baseline score 1, worst post-baseline score 0 | 0 | 0 | 0 | 0
  Baseline score 1, worst post-baseline score 1 | 1 | 1 | 1 | 5
  Baseline score 1, worst post-baseline score 2 | 0 | 0 | 0 | 0
  Baseline score 1, worst post-baseline score 3 | 0 | 0 | 0 | 0
  Baseline score 1, worst post-baseline score 4 | 0 | 0 | 0 | 0
  Baseline score 1, worst post-baseline score 5 | 0 | 0 | 0 | 0
  Baseline score 1, worst post-baseline score Missing | 0 | 0 | 0 | 0

19. Secondary Outcome: Part FE: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance: Baseline Score Versus (Vs) Worst Post-baseline Score
Description: as for outcome 17
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 404 Days)
Population: Safety Analysis Set included all participants who received at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 5
Participants
  Baseline score 0, worst post-baseline score 0 | 0 | 1
  Baseline score 0, worst post-baseline score 1 | 1 | 2
  Baseline score 0, worst post-baseline score 2 | 1 | 0
  Baseline score 0, worst post-baseline score 3 | 0 | 0
  Baseline score 0, worst post-baseline score 4 | 0 | 0
  Baseline score 0, worst post-baseline score 5 | 0 | 0
  Baseline score 0, worst post-baseline score Missing | 0 | 0
  Baseline score 1, worst post-baseline score 0 | 0 | 0
  Baseline score 1, worst post-baseline score 1 | 1 | 2
  Baseline score 1, worst post-baseline score 2 | 1 | 0
  Baseline score 1, worst post-baseline score 3 | 0 | 0
  Baseline score 1, worst post-baseline score 4 | 0 | 0
  Baseline score 1, worst post-baseline score 5 | 0 | 0
  Baseline score 1, worst post-baseline score Missing | 0 | 0

20. Secondary Outcome: Part A: Single Dose: Maximum Observed Plasma Concentration (Cmax) of M3814
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Day 1
Population: The PK Analysis Set included all participants who received at least one administration of M3814 and avelumab and had at least one measurable post-dose PK sample. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 10 | 4 | 6 | 4
nanogram per milliliter (ng/mL) | 392 (43.8) | 1030 (78.2) | 2340 (98.9) | 1710 (99.8) | 3190 (40.6)

21. Secondary Outcome: Part A: Multiple Dose: Maximum Observed Plasma Concentration (Cmax) of M3814
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Day 15
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 6 | 1 | 3 | 1
nanogram per milliliter (ng/mL) | 693 (131.1) | 2370 (38.8) | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values. | 2360 (33.6) | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values.

22. Secondary Outcome: Part B: Single Dose: Maximum Observed Drug Concentration (Cmax) of M3814
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 1, 2, 4 and 6 hour post-dose on Day 1
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 2 | 3 | 4 | 8
ng/mL | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values. | 1460 (19.0) | 854 (66.2) | 2380 (44.8)

23. Secondary Outcome: Part B: Multiple Dose: Maximum Observed Drug Concentration (Cmax) of M3814
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 1, 2, 4 and 6 hour post-dose on Day 10
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 2 | 3 | 4 | 6
ng/mL | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values. | 1220 (5.8) | 1420 (71.4) | 3150 (63.6)

24. Secondary Outcome: Part A: Single Dose: Time to Reach the Maximum Plasma Concentration (Tmax) of M3814
Description: Tmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Day 15
Population: PK Analysis Set included all participants who received at least 1 administration of peposertib and avelumab and had at least 1 measurable post-dose PK sample. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: hour
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 10 | 4 | 6 | 4
hour | 1.06 [1.00 to 1.12] | 2.02 [0.85 to 6.00] | 1.03 [0.87 to 2.08] | 1.51 [0.88 to 2.17] | 1.08 [1.00 to 2.05]

25. Secondary Outcome: Part A: Multiple Dose: Time to Reach the Maximum Plasma Concentration (Tmax) of M3814
Description: Tmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Day 15
Population: as for outcome 24
Measure: Median (Full Range); unit: hour
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 6 | 1 | 3 | 0
hour | 1.08 [1.00 to 2.98] | 1.16 [0.93 to 4.00] | NA [NA to NA] — Median and Full Range could not be calculated if fewer than 3 participants had reportable parameter values. | 1.87 [1.03 to 2.08] |

26. Secondary Outcome: Part B: Single Dose: Time to Reach the Maximum Plasma Concentration (Tmax) of M3814
Description: Tmax was obtained directly from the concentration versus time curve postdose.
Time Frame: Pre-dose, 2, 4 and 6 hours post-dose on Day 10
Population: as for outcome 24
Measure: Median (Full Range); unit: hour
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 2 | 3 | 4 | 9
hour | NA [NA to NA] — Median and Full range could not be calculated if fewer than 3 participants had reportable parameter values | 0.93 [0.85 to 1.00] | 1.42 [0.87 to 2.25] | 1.47 [0.72 to 3.82]

27. Secondary Outcome: Part B: Multiple Dose: Time to Reach the Maximum Plasma Concentration (Tmax) of M3814
Description: Tmax was obtained directly from the concentration versus time curve postdose.
Time Frame: Pre-dose, 2, 4 and 6 hours post-dose on Day 10
Population: as for outcome 24
Measure: Median (Full Range); unit: hour
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 3 | 3 | 3 | 6
hour | NA [NA to NA] — Median and Full Range could not be calculated if fewer than 3 participants had reportable parameter values. | 2.18 [1.98 to 2.78] | 2.28 [1.88 to 2.50] | 2.01 [1.85 to 5.03]

28. Secondary Outcome: Part A: Minimum Observed Drug Concentration (Cmin) of M3814
Description: Cmin is minimum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Day 1
Population: As described in the Statistical Analysis Plan Section 7 Changes to planned analyses, data for Cmin was not collected.
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: Part B: Minimum Observed Drug Concentration (Cmin) of M3814
Description: Cmin is minimum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 1, 2, 4 and 6 hour post-dose on Day 1
Population: As described in the Statistical Analysis Plan Section 7 Changes to planned analyses, data for Cmin was not collected.
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

30. Secondary Outcome: Part A: Average Plasma Concentration of M3814 Observed Post-dose (Cavg)
Description: Cavg is the average plasma concentration within 1 dosing interval obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Day 1
Population: As described in the Statistical Analysis Plan Section 7 Changes to planned analyses, data for Cavg was not collected.
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: Part B: Average Plasma Concentration of M3814 Observed Post-dose (Cavg)
Description: as for outcome 30
Time Frame: Pre-dose, 1, 2, 4 and 6 hour post-dose on Day 1
Population: As described in the Statistical Analysis Plan Section 7 Changes to planned analyses, data for Cavg was not collected.
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

32. Secondary Outcome: Part A: Fluctuation Index of M3814
Description: Fluctuation index is defined as percentage fluctuation (variation between maximum and minimum concentration at steady state), calculated as: 100*([Cmax Cmin]/Cavg).
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Day 1
Population: As described in the Statistical Analysis Plan Section 7 Changes to planned analyses, data for Fluctuation Index was not collected.
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

33. Secondary Outcome: Part B: Fluctuation Index of M3814
Description: as for outcome 32
Time Frame: Pre-dose, 1, 2, 4 and 6 hour post-dose on Day 1
Population: as for outcome 32
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

34. Secondary Outcome: Part A: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC0-t) of M3814
Description: Area under the serum concentration-time curve (AUC) from time zero to the last sampling time point at which the concentration is at or above lower limit of quantification (LLOQ).
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Day 1
Population: As described in the Statistical Analysis Plan Section 7 Changes to planned analyses, data for AUC0-t was not collected.
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

35. Secondary Outcome: Part B: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC0-t) of M3814
Description: as for outcome 34
Time Frame: Pre-dose, 1, 2, 4 and 6 hour post-dose on Day 1
Population: As described in the Statistical Analysis Plan Section 7 Changes to planned analyses, data for AUC0-t was not collected.
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

36. Secondary Outcome: Part A: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of M3814
Description: Area under the serum concentration-time curve from time zero to infinity (AUC0-inf). AUC0-inf calculated as AUC0-t + AUCextra. AUCextra represents the extrapolated part of AUC0-inf.
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Day 1
Population: As described in the Statistical Analysis Plan Section 7 Changes to planned analyses, data for AUC0-inf was not collected.
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

37. Secondary Outcome: Part B: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of M3814
Description: Area under the serum concentration-time curve from time zero to infinity (AUC0-inf). AUC0-infcalculated as AUC0-t + AUCextra.
Time Frame: Pre-dose, 1, 2, 4 and 6 hour post-dose on Day 1
Population: as for outcome 36
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

38. Secondary Outcome: Part A: Accumulation Ratio of Maximum Observed Drug Concentration [Racc(Cmax)] of M3814
Description: Accumulation ratio of Cmax was calculated as Cmax, after dosing on Day 15 divided by Cmax, after dosing on Day 1.
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Days 1 and 15
Population: PK Analysis Set included all participants who received at least 1 administration of peposertib and avelumab and had at least 1 measurable post-dose PK sample. Here, Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 5 | 1 | 3 | 0
ratio | 1.77 (95.1) | 1.47 (28.7) | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values. | 2.61 (45.0) |

39. Secondary Outcome: Part B: Accumulation Ratio of Cmax [Racc(Cmax)] of M3814
Description: Accumulation ratio of Cmax was calculated as Cmax, after dosing on Day 10 divided by Cmax, after dosing on Day 1.
Time Frame: Pre-dose, 1, 2, 4 and 6 hour post-dose on Day 1;Pre-dose, 2, 4 and 6 hours post-dose on Day 10
Population: as for outcome 38
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 1 | 3 | 3 | 6
ratio | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values. | 0.838 (24.8) | 2.15 (30.3) | 1.34 (39.3)

40. Secondary Outcome: Part A: Accumulation Ratio of AUC [Racc (AUC 0-12)] of M3814
Description: Accumulation ratio of AUC0-12 was calculated as AUC0-t, after dosing on Day 15 divided by AUC0-t, after dosing on Day 1.
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Days 1 and 15
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Groups:
- Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RTEdit: Participants received 100 milligrams (mg) of M3814 orally twice daily (BID) along with 800 mg of Avelumab once every 2 weeks (Q2W) from Day 1 until progressive disease (PD) or unacceptable toxicity.
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RTEdit | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 5 | 1 | 3 | 0
ratio | 2.36 (34.4) | 1.57 (74.0) | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values. | 4.32 (36.7) |

41. Secondary Outcome: Part B: Accumulation Ratio of AUC [Racc (AUC 0-24)] of M3814
Description: Accumulation ratio of AUC0-12 was calculated as AUC0-t, after dosing on Day 10 divided by AUC0-t, after dosing on Day 1.
Time Frame: Pre-dose, 1, 2, 4 and 6 hour post-dose on Day 1; Pre-dose, 2, 4 and 6 hours post-dose on Day 10
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 1 | 2 | 3 | 5
ratio | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values. | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values. | 1.44 (22.9) | 1.96 (25.6)

42. Secondary Outcome: Part A: Single Dose: Apparent Terminal Half-life (t1/2) of M3814
Description: T1/2 was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half. T1/2 was calculated by natural log 2 divided by Lambda z. Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Day 15
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 7 | 4 | 6 | 3
hour | 2.37 (17.9) | 3.94 (40.9) | 2.25 (27.4) | 5.24 (53.7) | 3.51 (35.5)

43. Secondary Outcome: Part A: Multiple Doses: Apparent Terminal Half-life (t1/2) of M3814
Description: as for outcome 42
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Day 15
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 5 | 1 | 3 | 0
hour | 5.60 (21.8) | 6.26 (158.4) | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values. | 11.4 (60.3) |

44. Secondary Outcome: Part B: Single Dose: Apparent Terminal Half-life (t1/2) of M3814
Description: as for outcome 42
Time Frame: Pre-dose, 1, 2, 4 and 6 hour post-dose on Day 1;Pre-dose, 2, 4 and 6 hours post-dose on Day 10
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 1 | 3 | 3 | 5
hour | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values. | 6.56 (30.4) | 6.95 (33.8) | 7.79 (39.3)

45. Secondary Outcome: Part B: Multiple Dose: Apparent Terminal Half-life (t1/2) of M3814
Description: as for outcome 42
Time Frame: Pre-dose, 1, 2, 4 and 6 hour post-dose on Day 1;Pre-dose, 2, 4 and 6 hours post-dose on Day 10
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 1 | 2 | 3 | 5
hour | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values. | NA (NA) — Geometric mean and Geometric mean coefficient of variation could not be calculated if fewer than 3 participants had reportable parameter values. | 7.50 (12.8) | 11.5 (38.2)

46. Secondary Outcome: Part A: Apparent Volume of Distribution During Terminal Phase (Vz/f) of M3814
Description: The apparent volume of distribution during the terminal phase following extravascular administration, based on the fraction of dose absorbed. Vz/f = Dose/(AUC0-inf multiplied by Lambda z).
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Day 1
Population: As described in the Statistical Analysis Plan Section 7 Changes to planned analyses, data for Vz/f was not collected.
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

47. Secondary Outcome: Part B: Apparent Volume of Distribution During Terminal Phase (Vz/f) of M3814
Description: as for outcome 46
Time Frame: Pre-dose, 1, 2, 4 and 6 hour post-dose on Day 1
Population: As described in the Statistical Analysis Plan Section 7 Changes to planned analyses, data for Vz/f was not collected.
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

48. Secondary Outcome: Part A: Apparent Clearance (CL/f) of M3814
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Day 1
Population: As described in the Statistical Analysis Plan Section 7 Changes to planned analyses, data for CL/f was not collected.
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

49. Secondary Outcome: Part B: Apparent Clearance (CL/f) of M3814
Description: as for outcome 48
Time Frame: Pre-dose, 1, 2, 4 and 6 hour post-dose on Day 1
Population: As described in the Statistical Analysis Plan Section 7 Changes to planned analyses, data for CL/f was not collected.
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

50. Secondary Outcome: Part A: Terminal Elimination Rate Constant (Lambda z) of M3814
Description: Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Day 1
Population: As described in the Statistical Analysis Plan Section 7 Changes to planned analyses, data for lambda z was not collected.
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

51. Secondary Outcome: Part B: Terminal Elimination Rate Constant (Lambda z) of M3814
Description: as for outcome 50
Time Frame: Pre-dose, 1, 2, 4 and 6 hour post-dose on Day 1
Population: as for outcome 50
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

52. Secondary Outcome: Part A: Number of Participants With Positive Antidrug Antibody (ADA)
Description: Blood samples were analyzed by a validated homogenous bridging electrochemiluminescence assay to detect the presence of antidrug antibodies (ADA). Number of participants with positive ADA were reported.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 516 Days)
Population: Safety Analysis Set included all participants who received at least 1 dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 11 | 4 | 6 | 4
Participants | 0 | 5 | 0 | 2 | 0

53. Secondary Outcome: Part B: Number of Participants With Positive Antidrug Antibody (ADA)
Description: as for outcome 52
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 513 Days)
Population: Safety Analysis Set included all participants who received at least 1 dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 3 | 3 | 4 | 9
Participants | 1 | 0 | 1 | 3

54. Secondary Outcome: Part FE: Number of Participants With Positive Antidrug Antibody (ADA)
Description: Serum samples were analyzed by a validated assay method to detect the presence of antidrug antibodies (ADA). Number of participants with positive ADA were reported.
Time Frame: Part FE: From the first study intervention to 508 days
Population: Safety Analysis Set included all participants who received at least 1 dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 5
Participants | 1 | 1

55. Secondary Outcome: Part A: Number of Participants With Confirmed Best Overall Response (BOR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: Confirmed BOR was defined as the percentage of participants who achieved confirmed complete responses (CR) or partial response (PR), according to RECIST version 1.1 assessed by the Investigator.CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Stable disease (SD)= Neither sufficient increase to qualify for progression of disease (PD) nor sufficient shrinkage to qualify for PR. PD: At least a 20 % increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. Confirmed CR=as at least two determinations of CR at least 4 weeks apart with no PD. Confirmed PR=as at least 2 determinations of PR or better (PR followed by PR or PR followed by CR), at least 4 weeks apart (not qualifying for a CR) with no PD in between. Percentage of Participants with confirmed BOR were reported.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 516 Days)
Population: Full Analysis Set included all participants who received at least 1 dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 11 | 4 | 6 | 4
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0
  Stable Disease or Non-CR/Non-PD | 2 | 1 | 1 | 0 | 1
  Progressive Disease | 2 | 7 | 0 | 2 | 1
  Not Evaluable | 0 | 3 | 3 | 4 | 2

56. Secondary Outcome: Part B: Number of Participants With Confirmed Best Overall Response (BOR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: as for outcome 55
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 513 Days)
Population: Full Analysis Set included all participants who received at least 1 dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 3 | 3 | 4 | 9
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0
  Stable Disease or Non-CR/Non-PD | 1 | 1 | 2 | 2
  Progressive Disease | 2 | 2 | 1 | 3
  Not Evaluable | 0 | 0 | 1 | 4

57. Secondary Outcome: Part FE: Number of Participants With Confirmed Best Overall Response (BOR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: as for outcome 55
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 404 Days)
Population: Full Analysis Set included all participants who receive at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 5
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 1
  Stable Disease or Non-CR/Non-PD | 2 | 1
  Progressive Disease | 1 | 1
  Not Evaluable | 1 | 2

58. Secondary Outcome: Part A: Duration of Response (DoR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator
Description: DOR was defined for participants with confirmed response, as the time from first documentation of objective response (Complete Response [CR] or Partial Response [PR]) to the date of first documentation of progression disease (PD) or death due to any cause, whichever occurred first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from first documentation of objective response until date of first documentation of PD or death due to any cause, whichever occurred first, assessed up to 516 Days
Population: Full Analysis Set: All participants who receive at least one dose of study intervention. Data could not be calculated as none of the participants showed objective response.
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

59. Secondary Outcome: Part B: Duration of Response (DoR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator
Description: as for outcome 58
Time Frame: Time from first documentation of objective response until date of first documentation of PD or death due to any cause, whichever occurred first, assessed up to 513 Days
Population: Full Analysis Set included all participants who receive at least one dose of study intervention. Data could not be calculated as none of the participants showed objective response.
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

60. Secondary Outcome: Part FE: Duration of Response (DoR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator
Description: as for outcome 58
Time Frame: Time from first documentation of objective response until date of first documentation of PD or death due to any cause, whichever occurred first, assessed up to 44 Weeks
Population: Full Analysis Set included all participants who receive at least one dose of study intervention. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 0 | 1
months |  | NA [NA to NA] — Median and Full range could not be calculated due to insufficient number of events.

61. Secondary Outcome: Part A: Progression-free Survival (PFS) Time According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) Assessed by Investigator
Description: Progression-Free Survival was calculated as the time from the start of any study intervention to the date of first documentation of objective progression of disease or death due to any cause, whichever occurs first. PD: At least a 20 percent (%) increase in the sum of the longest diameter (SLD) taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. The PFS was analyzed by using the Kaplan-Meier method.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 516 Days)
Population: Full Analysis Set included all participants who receive at least one dose of study intervention.
Measure: Median (Full Range); unit: months
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 11 | 4 | 6 | 4
months | 5.1 [1.87 to 13.77] | 1.9 [0.49 to 14.03] | 3.3 [0.03 to 3.68] | 1.8 [0.03 to 3.22] | 2.6 [0.03 to 2.89]

62. Secondary Outcome: Part B: Progression-free Survival (PFS) Time According to RECIST v 1.1 Assessed by Investigator
Description: as for outcome 61
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 513 Days)
Population: Full Analysis Set included all participants who receive at least one dose of study intervention.
Measure: Median (Full Range); unit: months
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 3 | 3 | 4 | 9
months | 1.9 [1.87 to 3.12] | 1.7 [1.68 to 8.34] | 3.4 [0.03 to 5.59] | 1.9 [0.03 to 5.55]

63. Secondary Outcome: Part FE: Progression-free Survival (PFS) Time According to RECIST v 1.1 Assessed by Investigator
Description: as for outcome 61
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 404 Days)
Population: Full Analysis Set included all participants who receive at least one dose of study intervention.
Measure: Median (Full Range); unit: months
Arm/Group | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 5
months | 2.7 [0.39 to 5.98] | 8.5 [0.69 to 8.51]

64. Secondary Outcome: Part A: Overall Survival
Description: Overall survival was defined as the time from treatment start to the date of death, regardless of the actual cause of the participant's death. The overall survival was analyzed by using the Kaplan-Meier method. Median, is estimated by Kaplan-Meier method which stands for the time that half of the participants are expected to be alive. Depending on the observed number of deaths, time of censoring for each participant, median survival time may not be reached or estimated (few deaths will lead the KM curve never crosses 50% survival line), hence median was not calculable for Part A: M3814 250 mg BID + Avelumab 800 mg Q2W arm. Participants that are still alive at the time of analysis will be censored and counted into the analysis.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 1359 Days)
Population: Full Analysis Set included all participants who receive at least one dose of study intervention. Here " Overall Number of Participants Analyzed" are equivalent to the number of participants who were evaluable for the outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 11 | 4 | 6 | 4
months | 25.5 [4.80 to 25.53] | 23.7 [0.92 to 23.7] | NA [0.76 to 7.13] — Median could not be calculated due to insufficient number of death, or the median survival is not reached yet | 3.4 [0.66 to 7.52] | 7.2 [2.73 to 7.23]

65. Secondary Outcome: Part B: Overall Survival
Description: Overall survival was defined as the time from treatment start to the date of death, regardless of the actual cause of the participant's death. The overall survival was analyzed by using the Kaplan-Meier method. Median, is estimated by Kaplan-Meier method which stands for the time that half of the participants are expected to be alive. Depending on the observed number of deaths, time of censoring for each participant, median survival time may not be reached or estimated (few deaths will lead the KM curve never crosses 50% survival line), hence median was not calculable for Part B of the study. Participants that are still alive at the time of analysis will be censored and counted into the analysis.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 1359 Days)
Population: as for outcome 64
Measure: Median (Full Range); unit: months
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 3 | 3 | 4 | 9
months | NA [4.01 to 9.00] — Median could not be calculated due to insufficient number of death or the median survival is not reached yet. | NA [3.4 to 19.38] — Median could not be calculated due to insufficient number of death or the median survival is not reached yet. | NA [6.60 to 18.69] — Median could not be calculated due to insufficient number of death or the median survival is not reached yet. | NA [1.08 to 7.98] — Median could not be calculated due to insufficient number of death or the median survival is not reached yet.

66. Secondary Outcome: Part FE: Overall Survival
Description: Overall survival was defined as the time from treatment start to the date of death, regardless of the actual cause of the participant's death. The overall survival was analyzed by using the Kaplan-Meier method. Participants that are still alive at the time of analysis will be censored and counted into the analysis.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 1359 Days)
Population: as for outcome 64
Measure: Median (Full Range); unit: months
Arm/Group | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 5
months | 6.4 [0.39 to 6.41] | 8.5 [0.69 to 9.66]

67. Secondary Outcome: Part A: Best Percent Change From Baseline in Tumor Size According to RECIST v 1.1
Description: Tumor size is derived as the best percent change from baseline in target lesions (sum of longest diameter for non-nodal lesions and short axis for nodal lesions) at each time point.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 516 Days)
Population: as for outcome 64
Measure: Median (Standard Deviation); unit: percent change
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 4 | 11 | 2 | 3 | 3
percent change | 15.8 (17.27) | 15.3 (15.38) | -4.5 (2.34) | 4.9 (8.07) | 13.6 (26.97)

68. Secondary Outcome: Part B: Best Percent Change From Baseline in Tumor Size According to RECIST v 1.1
Description: as for outcome 67
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 513 Days)
Population: as for outcome 64
Measure: Median (Standard Deviation); unit: percent change
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 3 | 3 | 3 | 5
percent change | 8.4 (19.59) | 0.3 (21.05) | -18.5 (8.19) | -0.7 (19.59)

69. Secondary Outcome: Part FE: Best Percent Change From Baseline in Tumor Size According to RECIST v 1.1
Description: as for outcome 67
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 404 Days)
Population: as for outcome 64
Measure: Median (Standard Deviation); unit: percent change
Arm/Group | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W
Number analyzed (Participants) | 3 | 4
percent change | 6.1 (14.98) | -13.3 (27.04)

70. Secondary Outcome: Part B: Number of Participants With Radiotherapy (RT)-Induced Toxicity According to NCI-CTCAE v 5.0
Description: Number of participants with radiotherapy-induced toxicities (mucositis and radiation dermatitis) were reported.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to 512.4 Days)
Population: Safety Analysis Set included all participants who received at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT
Number analyzed (Participants) | 3 | 3 | 4 | 9
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from first study intervention up to long term safety follow-up period (Up to 516 Days in Part A, Up to 513 days in Part B, Up to 404 days in Part FE); All-cause mortality was assessed up to 1359 days
Arm/Group | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W
All-Cause Mortality (participants affected / at risk) | 2/4 | 6/11 | 3/4 | 5/6 | 2/4 | 0/3 | 2/3 | 3/4 | 4/9 | 2/4 | 2/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 6/11 | 4/4 | 4/6 | 4/4 | 2/3 | 1/3 | 1/4 | 6/9 | 2/4 | 3/5
Other Adverse Events (participants affected / at risk) | 3/4 | 11/11 | 4/4 | 6/6 | 4/4 | 3/3 | 3/3 | 4/4 | 9/9 | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W (N=4) | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W (N=11) | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W (N=4) | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W (N=6) | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W (N=4) | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT (N=3) | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT (N=3) | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT (N=4) | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT (N=9) | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W (N=4) | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W (N=5)
Anaemia (Blood and lymphatic system disorders) | NA | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | NA | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | NA | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | NA | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | NA | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | NA | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | NA | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: M3814 100 mg BID + Avelumab 800 mg Q2W (N=4) | Part A: M3814 200 mg BID + Avelumab 800 mg Q2W (N=11) | Part A: M3814 250 mg BID + Avelumab 800 mg Q2W (N=4) | Part A: M3814 300 mg BID + Avelumab 800 mg Q2W (N=6) | Part A: M3814 400 mg BID + Avelumab 800 mg Q2W (N=4) | Part B: M3814 100 mg BID + Avelumab 800 mg Q2W + RT (N=3) | Part B: M3814 150 mg BID +Avelumab 800 mg Q2W + RT (N=3) | Part B: M3814 200 mg BID + Avelumab 800 mg Q2W + RT (N=4) | Part B: M3814 250 mg BID + Avelumab 800 mg Q2W + RT (N=9) | Part Food Effect: M3814 100 mg BID + Avelumab 800 mg Q2W (N=4) | Part Food Effect: M3814 200 mg BID + Avelumab 800 mg Q2W (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual field defect (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 7 (8) | 3 (4) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 7 (9) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 6 (7) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 5 (6) | 1 (1) | 4 (5)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (4)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 2 (2)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Blood phosphorus increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Data collection and analysis of Pharmacokinetics and Immunogenicity for Avelumab were omitted and not conducted due to business reason. PK parameters for avelumab were planned but the decision was made to only list and summarize with descriptive statistics avelumab concentrations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-11-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT03724890/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT03724890/SAP_001.pdf